CLINICAL TRIAL: NCT06691841
Title: Effect of Chlorhexidine Gluconate in Oral Care of Patients With Endotracheal Intubation Based on 16sRNA Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Sheng Wang MD PhD, director, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22K204
Record Dates: First submitted 2022-09-23; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-09

CONDITIONS: Intubation, Endotracheal; Oral Hygiene
Keywords: Chlorhexidine Gluconate; Endotracheal Intubation; 16sRNA
MeSH Terms: interventions — chlorhexidine gluconate; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normal Saline Group (Other): oral wiping and oral care solution rinsing, oral care solution was 0.9% normal saline, and oral care frequency was 3 times a day.
  Interventions: Other: normal saline
- Chlorhexidine group (Experimental): oral wiping and oral care solution rinsing, oral care solution was 0.12% Chlorhexidine gluconate solution, and oral care frequency was 3 times a day.
  Interventions: Drug: Chlorhexidine Gluconate

INTERVENTIONS:
Drug: Chlorhexidine Gluconate — oral wiping and oral care solution rinsing, oral care solution was 0.12% chlorhexidine gluconate, and the frequency of oral care was 3 times a day.
  Other Names: jinkouxin
  Arms: Chlorhexidine group
Other: normal saline — oral wiping and oral care solution rinsing, oral care solution was 0.9% normal saline, and the frequency of oral care was 3 times a day.
  Arms: Normal Saline Group

SUMMARY:
Evaluation of the application effect of compound chlorhexidine gargle in oral care of patients with endotracheal intubation based on 16s RNA technology.

DETAILED DESCRIPTION:
Evaluation of the application effect of compound chlorhexidine gargle in oral care of patients with endotracheal intubation based on 16s RNA technology. Between September 2022 and March 2023, 68 patients admitted to the ICU for endotracheal intubation were collected. They were randomly divided into intervention group and control group, with 34 cases in each group. The control group used the method of wiping, washing and saline (0.9%) three times a day, and the intervention group was using the method of wiping, washing and 0.12% chlorhexidine gluconate three times a day.The results were analyzed at three time points before the first oral care after intubation, before oral care 48 hours after intubation, and before oral care on the 5th day after intubation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years; ② Complete clinical data; ③ Expected duration of orotracheal intubation for mechanical ventilation exceeding 5 days.

Exclusion Criteria:

* Patients with abnormal coagulation function, severe respiratory burns, oral surgery, lung and systemic infections; ② Patients expected to die within 48 hours after extubation; ③ Patients with actual duration of orotracheal intubation for mechanical ventilation less than 5 days.

Exclusion During Study:

* Failure to follow the prescribed plan; ② Incomplete data; ③ Patients who voluntarily withdraw from treatment during the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Changes in the oral microbiota | Immediately after enrollment; 48 hrs after intubation；5 days after intubation
  objective analysis results based on 16s RNA technology

SECONDARY OUTCOMES:
oral complications | mechanical ventilation at 0 hours, 2 days, and 5 days post-intervention
  Oral complication occurrences: The occurrences of oral mucosa bleeding, oral inflammation, oral ulcers, fungal and herpes virus infections, tongue falling backwards, laryngeal edema, granulomas, and other complications were recorded in elderly patients undergoing mechanical ventilation at 0 hours, 2 days, and 5 days post-intervention. Diagnosis was confirmed through blood routine tests, histopathological examinations, smear tests, fungal cultures, or other methods.
plaque Index | mechanical ventilation at 0 hours, 2 days, and 5 days post-intervention
  Dental Plaque Index: The mesial buccal, middle buccal, distal buccal, and lingual surfaces of the teeth in elderly patients undergoing mechanical ventilation were examined and scored using a combination of visual inspection and probing. A score of 0 indicates no plaque at the gingival margin, 1 indicates a thin layer of plaque at the gingival margin, 2 indicates moderate plaque at the gingival margin or interproximal area, and 3 indicates abundant soft debris within the gingival sulcus, at the gingival margin, and in the interproximal area. The Dental Plaque Index is calculated as the sum of the plaque scores for each tooth divided by the total number of teeth examined.
whether VAP occurs | Immediately after enrollment; 48 hrs after intubation；5 days after intubation
  the recorder records whether VAP occurs after endotracheal intubation;Ventilator-associated pneumonia (VAP) refers to pneumonia that occurs between 48 hours after the initiation of mechanical ventilation (MV) and 48 hours after extubation. It is an important type of hospital-acquired pneumonia (HAP). Among them, pneumonia that occurs within 4 days of MV is classified as early-onset VAP, while that occurring on or after the 5th day is classified as late-onset VAP.
28-day mortality rate | 28 days post-randomization
  Survival status at day 28

CONTACTS AND LOCATIONS:
Overall Officials: sheng wang, PHD, Study Director — Shanghai Tenth People's Hospital, Tongji University School of Medicine, Shanghai, China
Locations (1):
- Changcui Qiu, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Qiu C, Tang L, Hang Z, Wei K, Wang S, Zhu X, Wang Q. Effect of chlorhexidine vs. saline for oral care on oral microbiota and prognosis of elderly mechanically ventilated patients in the intensive care unit: a single-center, single-blind, randomized controlled trial. BMC Oral Health. 2025 Dec 28. doi: 10.1186/s12903-025-07579-7. Online ahead of print. PMID 41456054